CLINICAL TRIAL: NCT06023602
Title: Effectiveness of Generic Cetrorelix Acetate Versus Reference Cetrorelix Acetate for Ovarian Stimulation Using a GnRH Antagonist Protocol in Women Undergoing IVF: A Multicenter Non-inferiority, Randomised Controlled Trial
Brief Title: Effectiveness of Generic Versus Reference Cetrorelix Acetate for Ovarian Stimulation Using a Gonadotropin-releasing Hormone（GnRH）Antagonist Protocol in Women Undergoing IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Principal Investigator, He Cai, Principal Investigator, Northwest Women's and Children's Hospital, Xi'an, Shaanxi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-038
Record Dates: First submitted 2023-08-18; First posted 2023-09-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Generic cetrorelix acetate (Experimental)
  Interventions: Drug: Generic cetrorelix acetate
- Reference cetrorelix acetate (Active Comparator)
  Interventions: Drug: Reference cetrorelix acetate

INTERVENTIONS:
Drug: Generic cetrorelix acetate — Generic cetrorelix acetate (0.25 mg SC)
  Arms: Generic cetrorelix acetate
Drug: Reference cetrorelix acetate — reference cetrorelix acetate (0.25 mg SC)
  Arms: Reference cetrorelix acetate

SUMMARY:
The goal of this clinical trial is to compare the clinical outcomes using different cetrorelix acetate in the context of a GnRH antagonist protocol for ovarian stimulation in women undergoing IVF or intracytoplasmic sperm injection(ICSI) treatment.The main question it aims to answer is whether the generic cetrorelix acetate is non-inferior to the reference product in the GnRH antagonist based protocol for women undergoing IVF. Ovarian stimulation was achieved by several types of follicle-stimulating hormone(FSH) or by FSH combined with luteinizing hormone activity. Daily dose of generic cetrorelix acetate (0.25 mg SC) or original cetrorelix acetate (0.25 mg SC) will be administered when the lead follicle was 14 mm. When more than two follicles reached 17 mm, oocyte maturation was triggered with 250 mcg of recombinant human chorionic gonadotropin.

ELIGIBILITY:
Inclusion Criteria:

* Infertile couples plan to undergo IVF / ICSI pregnancy treatment into screening procedures and clinical study

  1. All subjects should sign the informed consent form
  2. Infertile women <43 years old
  3. With flexible GnRH antagonist

Exclusion Criteria:

* Subjects could not enter the study if they meet any one of the following criteria

  1. Preimplantation Genetic Testing (PGT)
  2. Untreated hydrosalpinges, moderate or severe endometriosis, recurrent spontaneous miscarriage, endometrial pathology, uterine malformations, etc
  3. Endocrine diseases (such as hyperthyroidism, hyperprolactinemia, etc.) or other systemic disease and other systemic diseases (such as hypertension, diabetes, etc.)．
  4. Other factors were considered inappropriate by the investigator to participate, or assisted reproductive technology/pregnancy contraindications

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1338 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | Through study completion, an average of 18 months
  For the first live birth (gestation≥ 24 weeks) in one in vitro fertilization/intracytoplasmic sperm injection egg retrieval cycle (fresh and frozen-thawed embryo transfer cycle)

CONTACTS AND LOCATIONS:
Locations (1):
- He Cai, Xi'an, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dovey S, McIntyre K, Jacobson D, Catov J, Wakim A. Is a premature rise in luteinizing hormone in the absence of increased progesterone levels detrimental to pregnancy outcome in GnRH antagonist in vitro fertilization cycles. Fertil Steril. 2011 Sep;96(3):585-9. doi: 10.1016/j.fertnstert.2011.06.042. Epub 2011 Jul 20. PMID 21774931
- [Background] Liu X, Wen W, Wang T, Tian L, Li N, Sun T, Wang T, Zhou H, Zhang N, Qu P, Mol BW, Li W, Shi J. Increased versus standard gonadotrophin dosing in predicted poor responders of IVF: an open-label randomized controlled trial. Hum Reprod. 2022 Jul 30;37(8):1806-1815. doi: 10.1093/humrep/deac113. PMID 35595197